CLINICAL TRIAL: NCT04684732
Title: Relationship Between Renal Function and Pharmacokinetics of Apixaban and Clinical Outcome of Apixaban in Thai Non-valvular Atrial Fibrillation Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Chulalongkorn University (Other)
Collaborators: Thammasat University (Other)
Responsible Party: Principal Investigator, Pheeraphat Sarppreuttikun, Principle Investigator, Chulalongkorn University
Other Study IDs: 632/63
Record Dates: First submitted 2020-12-14; First posted 2020-12-24 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Atrial Fibrillation
Keywords: Apixaban; Pharmacokinetic; Pharmacodynamic; Cardioembolic stroke; Ischemic stroke
MeSH Terms: conditions — Atrial Fibrillation; Embolic Stroke; Ischemic Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Apixaban dose concordant to leaflet: Patients who were prescribed apixaban dose concordant to apixaban leaflet approved by Thai FDA
- Apixaban dose discordant to leaflet: Patients who were prescribed apixaban dose discordant to apixaban leaflet approved by Thai FDA

SUMMARY:
The purpose of this study is to assess pharmacokinetics and pharmacodynamics of Apixaban and clinical outcome of Apixaban in Thai patients with nonvalvular atrial fibrillation with varying degree of creatinine clearance

DETAILED DESCRIPTION:
This study is divided into two parts.

The first part is a multiple dose pharmacokinetic and pharmacodynamics study of Apixaban in patient with stable renal function. The primary purpose of this study is to provide a clear understanding of the effect of creatinine clearance on pharmacokinetics and pharmacodynamics of Apixaban among Thai patients with nonvalvular atrial fibrillation. To assess the pharmacokinetics and pharmacodynamics of Apixaban, This study will enroll 30 subjects who meet the inclusion criteria.

The second part of this study will retrospectively determine the occurrent of clinical outcome between patients who were prescribed apixaban dose concordant and discordant to the drug leaflet. A total of 241 subjects will be recruited. The follow up period will begin from the time of initiation of apixaban until occurrent of stoke, transient ischemic attack, systemic embolism, bleeding, or death.

ELIGIBILITY:
Part I

Inclusion Criteria:

* Patients with nonvalvular atrial fibrillation
* Patients who is receiving a stable dose of apixaban for primary or secondary prevention of stroke, transient ischemic attack, and systemic embolism.

Exclusion Criteria:

* Pregnant or lactating
* End stage renal disease patients who required chronic renal replacement therapy to sustained life
* History of acute kidney injury within the previous 3 months
* Severe hepatic impairment (Child-Pugh class C)
* Any gastrointestinal disorder that could impact the absorption of study drug
* CYP3A4 Moderate/Strong Inhibitors: ketoconazole, itraconazole, voriconazole, posaconazole, ritonavir, naproxen, clarithromycin, rifampicin, phenytoin, carbamazepine, phenobarbital, diltiazem, and St.John's Wort

Part II

Inclusion Criteria:

* Patients with nonvalvular atrial fibrillation
* Patients who was prescribed apixaban for primary or secondary prevention of stroke, transient ischemic attack, and systemic embolism.

Exclusion Criteria:

* Pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thai patients with nonvalvular atrial fibrillation receiving a stable dose of apixaban for primary or secondary prevention of stroke, transient ischemic attack, or systemic embolism.
Sampling Method: Non-Probability Sample
Enrollment: 241 (Estimated)
Dates: Start 2020-12-14 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Steady state area under the concentration-time curve from pre-dose to 12 hours post-dose (AUC(0-12)) of Apixaban | pre-dose to 12 hours post-dose
  AUC(0-12) is measured by plasma concentration of apixaban over time. The mean are reported in nanogram hours per milliliter (ng*h/mL).

SECONDARY OUTCOMES:
Number of participants with first event of stroke, transient ischemic attack, systemic embolism (SE), or all-cause death during the follow up period | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed until July 31, 2020
  Diagnosis of stroke is defined as the nontraumatic focal neurological deficit lasting at least 24 hours, and includes ischemic stroke, hemorrhagic stroke, ischemic stroke with hemorrhagic conversion, stroke of uncertain type, and retinal ischemic event (embolism, infarction). Diagnosis of SE is defined as a clinical history consistent with an acute loss of blood flow to a peripheral artery (or arteries), supported by evidence of embolism from surgical specimens, autopsy, angiography, vascular imaging, or other objective testing.
Number of patients with event of major or nonmajor (International Society on Thrombosis and Hemostasis [ISTH]) bleeding during the follow up period | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed until July 31, 2020
  ISTH major bleeding criteria is defined as a bleeding event that was: clinically overt bleeding accompanied by a decrease in hemoglobin (Hgb) of 2 g/dL or more, and/or a transfusion of 2 or more units of packed red blood cells; bleeding that occurred in at least 1 of the following critical sites: intracranial, intraspinal, intraocular (within the corpus of the eye; a conjunctival bleed is not an intraocular bleed), pericardial, intra-articular, intramuscular with compartment syndrome, and retroperitoneal; bleeding that was fatal.
  ISTH nonmajor bleeding is defined as clinically overt, that satisfies none of the additional criteria required for the event to be adjudicated as a major bleeding event, that led to either hospital admission for bleeding, physician-guided medical or surgical treatment for bleeding, or a change in antithrombotic therapy.

OTHER OUTCOMES:
Steady-state maximum observed plasma concentration of Apixaban | pre-dose to 12 hours post-dose
  Maximum observed drug concentration in plasma after administration (Cmax) of apixaban at steady-state
Steady-state minimum observed plasma concentration of Apixaban | pre-dose to 12 hours post-dose
  Minimum observed drug concentration in plasma after administration (Cmin) of apixaban at steady-state
Steady state elimination of half-life of Apixaban | pre-dose to 12 hours post-dose
  Mean terminal phase plasma t½ of apixaban at steady-state
Steady state Anti-Xa activity | pre-dose to 12 hours post-dose
  Anti-Xa activity will be measured by chromogenic anti-Xa activity assay

CONTACTS AND LOCATIONS:
Locations (1):
- King Chulalongkorn Memorial Hospital, Pathum Wan, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No